CLINICAL TRIAL: NCT06085365
Title: A Multicenter, Open-label, Parallel Controlled, Prospective Cohort Study Evaluating Immunonutrition on the Improvement of Postoperative Adjuvant Chemotherapy Related Adverse Reactions in Patients With Gastrointestinal Tumors
Brief Title: Effects of Immunonutrition on the Improvement of Postoperative Adjuvant Chemotherapy Related Adverse Reactions in Patients With Gastrointestinal Tumors
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Yunpeng Liu, Clinical Professor, China Medical University, China
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CLOG2301
Record Dates: First submitted 2023-09-30; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Gastrointestinal Tumors; Immunonutrition; Postoperative Adjuvant Chemotherapy
MeSH Terms: conditions — Digestive System Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (Placebo Comparator): normal diet group
  Interventions: Drug: fluorouracil based chemotherapy regimens
- Immunonutrition Group (Experimental): Immunonutrition (Suyusu) 250ml oral twice one day d1-d21 for two cycles
  Interventions: Drug: Immunonutrition （Su yusu); Drug: fluorouracil based chemotherapy regimens

INTERVENTIONS:
Drug: Immunonutrition （Su yusu) — Immunonutrition （Su yusu） 250ml oral twice a day d1-d21
  Arms: Immunonutrition Group
Drug: fluorouracil based chemotherapy regimens — fluorouracil based chemotherapy regimens

SUMMARY:
Evaluate the effects of Suyusu (immunonutrition) in postoperative adjuvant chemotherapy for gastrointestinal cancer patients. The main endpoint of the study was the incidence of chemotherapy related adverse reactions (including bone marrow suppression, nausea and vomiting, diarrhea, and mucositis) in patients after two cycles of chemotherapy. The secondary endpoint indicators were: quality of life score (EORTC-QLQ-C30), nutritional risk score (PG-SGA, NRS2002), nutritional assessment indicators, changes in immune microenvironment, analysis of psychological status, survival time (1-year progression free survival rate), treatment tolerance (dose intensity, rate of treatment interruption, delay), etc.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily and sign an informed consent form;
2. Age ≥ 18 years old and ≤ 75 years old;
3. Patients with stage II-III gastrointestinal malignancies with clear pathological diagnosis and undergoing radical surgery
4. No adjuvant chemotherapy received after surgery
5. The Eastern Cancer Collaborative Group's Physical State Score (ECOG) is 0-2 points;
6. No contraindications to chemotherapy and the use of fluorouracil based chemotherapy regimens;

Exclusion Criteria:

1. Allergy to the components of immune nutrients, allergic constitution, or other inability to eat;
2. Participated in other drug or food clinical trials within 2 months prior to enrollment;
3. Having a history of immune deficiency, including HIV testing positive, or having other acquired or congenital immune deficiency diseases, or having a history of organ transplantation, or active infections that are not suitable for chemotherapy (as determined by the researcher);
4. Subjects cannot guarantee compliance after participating in the study;
5. Other researchers believe that it is not suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2023-07-24 (Actual); Primary Completion 2024-07-24 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of chemotherapy related adverse reactions | the first two cycles of chemotherapy. (each cycle is 21 ± 3 days)
  including bone marrow suppression, nausea and vomiting, diarrhea, and mucositis and so on.

SECONDARY OUTCOMES:
quality of life score | the first two cycles of chemotherapy. (each cycle is 21 ± 3 days)
  EORTC(The European Organization for Reasearch and Treatment of Cancer)-QOL-C30 (Quality of Life Questionnare-Core 30), patients need to answer all the questions by circling the number (1,2,3,4), big number means the worse quality of life score
nutritional risk score | the first two cycles of chemotherapy. (each cycle is 21 days)
  (PG-SGA) the patient-generated subjective global assessment. The result (A means well-nourished, B means middling-cacotrophia, C means severe malnutrition). Nutritional risk Screening Form 2002 (NRS2002), score ≥3 means patients with nutritional risk, score <3 patients with no nutritional risk. We use the two methods to evaluate the nutritional risk score.
changes in immune microenvironment | the first two cycles of chemotherapy. (each cycle is 21 ± 3 days)
  cytokines (pg/ml)
survival time | 1-year
  1-year progression free survival rate
treatment tolerance | the first two cycles of chemotherapy. (each cycle is 21 ± 3 days)
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
changes in immune microenvironment | the first two cycles of chemotherapy. (each cycle is 21 ± 3 days)
  Intestinal flora changes

CONTACTS AND LOCATIONS:
Locations (1):
- The First Hospital of China Medical University, Shenyang, Liaoning, China